CLINICAL TRIAL: NCT03714490
Title: MRI Simulation-guided Boost in Short-course Preoperative Radiotherapy (SCPRT) Followed by Consolidation Chemotherapy Versus Long Course Chemoradiation for Unresectable Rectal Cancer
Brief Title: MRI Simulation-guided Boost in Short-course Preoperative Radiotherapy for Unresectable Rectal Cancer
Acronym: SUNRISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, JIN JING, Professor, Director of medical services, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC201807007
Record Dates: First submitted 2018-10-09; First posted 2018-10-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Rectal Neoplasms
Keywords: rectal cancer; short-term radiotherapy; neoadjuvant chemotherapy; total mesorectal excision; MRI-simulation; boost
MeSH Terms: conditions — Rectal Neoplasms | interventions — XELOX

STUDY DESIGN:
Intervention Model Description: Randomized phase II trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention of Experimental group includes: Radiotherapy, followed by chemotherapy with capecitabine, oxaliplatin, and then surgery. The detail of procedure: 1, short-course preoperative radiotherapy(SCPRT) , which consists of SCPRT, 5 Gray(Gy) x 5, 4Gy for boost on the gross tumour volume(GTV) with MRI-simulation alone; 2,then after 7-10 days of radiotherapy completed, patients will receive consolidation chemotherapy, given in 3 week cycle of capecitabine 1000 mg/m2 twice daily, day 1-14 combined with oxaliplatin 130 mg/m2 once. In total, 4 cycles of neoadjuvant chemotherapy are prescribed preoperatively, then followed by a total mesorectal excision(TME) and postoperative adjuvant chemotherapy.
  Interventions: Radiation: SCPRT; Drug: CAPOX
- Control group (Active Comparator): The intervention of Control group includes:Radiotherapy, capecitabine, and surgery. The detail of procedure: 1, long-term chemoradiotherapy(CRT), which consists of a long-term chemoradiation (2 Gy x 25 with capecitabine) preoperatively; 2, 6-8 weeks after chemoradiation, total mesorectal excision(TME) and then postoperative adjuvant chemotherapy. The radiotherapy is given in combination with capecitabine in a dose of 825 mg/m2 twice daily on days when radiotherapy, excluding weekends.
  Interventions: Radiation: CRT

INTERVENTIONS:
Radiation: SCPRT — Short-course preoperative radiotherapy(SCPRT), which consists of 5 Gy x 5f and 4Gy for boost on the GTV with MRI-simulation alone.
  Arms: Experimental group
Radiation: CRT — Long-term chemoradiotherapy(CRT), which consists of a long-term chemoradiation (2 Gy x 25 with capecitabine) preoperatively.
  Arms: Control group
Drug: CAPOX — Patients will receive consolidation chemotherapy after 7-10 days of SCPRT completed, given in 3 week cycle of capecitabine 1000 mg/m2 twice daily, day 1-14 combined with oxaliplatin 130 mg/m2 once. In total, 4 cycles of neoadjuvant chemotherapy are scheduled before surgery.
  Other Names: capecitabine, oxaliplatin
  Arms: Experimental group

SUMMARY:
Improvements in downstaging are required when using preoperative chemoradiation for unresectable rectal cancer. There is therefore a need to explore more effective schedules. The study arm will receive MRI simulation-guided boost in short-course preoperative radiotherapy followed by consolidation chemotherapy , which may enhance the shrinkage of tumor comparing with the concurrent chemoradiation.

DETAILED DESCRIPTION:
The study is a prospective phase II randomized multicenter trial. The purpose of this study is to compare short-term radiotherapy with MRI simulation-guided boost followed by consolidation chemotherapy(Experimental group) with preoperative long-term chemoradiotherapy(Control group) for middle-lower unresectable locally advanced rectal cancer evaluated by MRI. The primary endpoint is the rate of R0 resection and cCR, and the secondary objectives are local recurrence-free survival, distant metastasis-free survival, disease-free survival and overall survival at 3-year and 5-year follow up. Furthermore, pathological complete response rate, the acute and late toxicity profile and quality of life (QOL) after 3 years follow-up are secondary endpoints. The exploratory end point includes the circulating tumor DNA, and other potential biomarkers from tumor tissue and blood sample for treatment response and survival predicting. For each group, a plan for collection of serum/plasma/feces at baseline and different stages during or after treatment and for obtaining fresh tumor tissue for freezing prior to treatment was defined in the protocol.

The SUNRISE-trial has been designed by National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences, Peking Union Medical College, and the hypothesis is R0 resection rate in Experimental group was superior to that in Control group.

Interim analysis design: As a phase II trial, the safety of experimental intervention is a major concern. We took the toxicity data from STELLAR, a phase III randomized study led by our center, as a reference. The incidence of G3 and above side effects in the short course radiotherapy with sequential neoadjuvant chemotherapy group was 28%, and that in the standard long-course concurrent chemoradiotherapy control group was 5%. Considering that boost dose may increase toxicity, if severe toxicity in the study group significantly exceeds that in the control group by more than 35%, it is up to the principal investigator to decide whether to modify the study protocol or terminate the study. The sample size of the interim analysis was calculated by the Z-pooled test, with α=0.05 (one-sided test), 1-β=0.90, using PASS 11 software. The frequency of the toxicity of G3 and above should be compared when neoadjuvant therapy was completed in 21 patients enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven rectal adenocarcinoma;
* Distance between tumour and anal verge≤ 10cm;
* Locally advanced tumour;(AJCC Cancer Staging:T3, T4 or N+)
* Mesorectal fascia(MRF)+ or T4b evaluated by pelvic MRI;
* Eastern Cooperative Oncology Group(ECOG) performance score ≤ 1;
* Written informed consent;
* Mentally and physically fit for chemotherapy;
* Adequate blood counts: White blood cell count ≥3.5 x 109/L Haemoglobin levels ≥100g/L Platelet count ≥100 x 109/L Creatinine levels ≤1.0× upper normal limit（UNL） Urea nitrogen levels ≤1.0× upper normal limit（UNL） Alanine aminotransferase(ALT) ≤1.5× upper normal limit（UNL） Aspartate aminotransferase(AST) ≤1.5× upper normal limit（UNL） Alkaline phosphatase(ALP) ≤1.5× upper normal limit（UNL） Total bilirubin(TBIL) ≤1.5× upper normal limit（UNL）
* No excision of tumor, chemotherapy or other anti-tumor treatment after the diagnosis.

Exclusion Criteria:

* Distant metastases;
* Recurrent rectal cancer;
* Active Crohn's disease or ulcerative colitis;
* Concomitant malignancies;(except basocellular carcinoma or in-situ cervical carcinoma)
* Allergic to Fluorouracil or Platinum drugs;
* Contraindications to MRI for any reason;
* Concurrent uncontrolled medical condition;
* Pregnancy or breast feeding;
* Known malabsorption syndromes or lack of physical integrity of upper gastrointestinal tract;
* Symptoms or history of peripheral neuropathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-23 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
R0(microscopically margin-negative) resection and cCR rate | 1-month after surgery completed
  The composite outcome of R0 (microscopically margin-negative) resection and cCR, that is, the combined rate of radical resection and cCR management after neoadjuvant treatment.

SECONDARY OUTCOMES:
local recurrence-free survival | 3-year and 5-year
  the time from surgery to local recurrence
distant metastasis-free survival | 3-year and 5-year
  the time from diagnosis to metastasis
disease-free survival | 3-year and 5-year
  the time from surgery to recurrence
overall survival | 3-year and 5-year
  the time from diagnosis to death
pathological complete response rate | 1-month after surgery completed
  pathological complete response in surgery specimen
clinical complete response rate | 3-month after neoadjuvant treatment
  clinical complete response evaluated by MDT
the acute toxicity profile | 1-month
  the frequency of acute adverse events during and after treatment in 1-month, including gastrointestinal (vomiting, diarrhea and incontinence), dermatitis, and hematologic toxicity evaluated weekly by the Common Terminology Criteria 4.0.
the late toxicity profile | 3-year
  the late toxicity after treatment completion for 1-month, the frequency of late adverse events after 1-month of treatment, including gastrointestinal function, fistula, and hematologic toxicity, evaluated regularly by LENT-SOMA scoring systems.
general quality of life (QoL) by QLQ-30 | 3-year
  general quality of life of patients evaluated by questionaire of EORTC QLQ-C30. The higher score in total indicates the worse quality of life in general.
QoL by QLO-CR29 | 3-year
  quality of life related to colorectal disease of patients evaluated by questionaire of EORTC QLQ-CR29. The higher score in total of this module indicates the worse quality of life by colorectal module.
Sum of sustained clinical complete response rate and R0 resection rate | 12 months after neoadjuvant therapy
  the rate of sustained clinical complete response plus rate of R0 resection

OTHER OUTCOMES:
circulating tumor DNA, single cells, Cytokines and other potential biomarkers such as T-cell receptor | 3-year
  The exploratory end point for predicting of treatment response and survival. The circulating tumor DNA test by sequencing will includes KRAS, NRAS, BRAF,PI3K,TP53,PTEN, EGFR, NEGF etc (509-gene panel). And Measuring change in T cell receptor sub-types during treatment.Single cells test by cytof. Cytokines test by the Olink Proteomics panel.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, M.D., Study Director — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] Chen W, Zheng R, Zeng H, Zhang S, He J. Annual report on status of cancer in China, 2011. Chin J Cancer Res. 2015 Feb;27(1):2-12. doi: 10.3978/j.issn.1000-9604.2015.01.06. PMID 25717220
- [Background] Glynne-Jones R, Wyrwicz L, Tiret E, Brown G, Rodel C, Cervantes A, Arnold D; ESMO Guidelines Committee. Rectal cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2017 Jul 1;28(suppl_4):iv22-iv40. doi: 10.1093/annonc/mdx224. No abstract available. PMID 28881920
- [Background] Bujko K, Wyrwicz L, Rutkowski A, Malinowska M, Pietrzak L, Krynski J, Michalski W, Oledzki J, Kusnierz J, Zajac L, Bednarczyk M, Szczepkowski M, Tarnowski W, Kosakowska E, Zwolinski J, Winiarek M, Wisniowska K, Partycki M, Beczkowska K, Polkowski W, Stylinski R, Wierzbicki R, Bury P, Jankiewicz M, Paprota K, Lewicka M, Cisel B, Skorzewska M, Mielko J, Bebenek M, Maciejczyk A, Kapturkiewicz B, Dybko A, Hajac L, Wojnar A, Lesniak T, Zygulska J, Jantner D, Chudyba E, Zegarski W, Las-Jankowska M, Jankowski M, Kolodziejski L, Radkowski A, Zelazowska-Omiotek U, Czeremszynska B, Kepka L, Kolb-Sielecki J, Toczko Z, Fedorowicz Z, Dziki A, Danek A, Nawrocki G, Sopylo R, Markiewicz W, Kedzierawski P, Wydmanski J; Polish Colorectal Study Group. Long-course oxaliplatin-based preoperative chemoradiation versus 5 x 5 Gy and consolidation chemotherapy for cT4 or fixed cT3 rectal cancer: results of a randomized phase III study. Ann Oncol. 2016 May;27(5):834-42. doi: 10.1093/annonc/mdw062. Epub 2016 Feb 15. PMID 26884592
- [Background] Braendengen M, Tveit KM, Berglund A, Birkemeyer E, Frykholm G, Pahlman L, Wiig JN, Bystrom P, Bujko K, Glimelius B. Randomized phase III study comparing preoperative radiotherapy with chemoradiotherapy in nonresectable rectal cancer. J Clin Oncol. 2008 Aug 1;26(22):3687-94. doi: 10.1200/JCO.2007.15.3858. PMID 18669453
- [Background] Burbach JP, den Harder AM, Intven M, van Vulpen M, Verkooijen HM, Reerink O. Impact of radiotherapy boost on pathological complete response in patients with locally advanced rectal cancer: a systematic review and meta-analysis. Radiother Oncol. 2014 Oct;113(1):1-9. doi: 10.1016/j.radonc.2014.08.035. Epub 2014 Oct 1. PMID 25281582
- [Background] Teo MTW, McParland L, Appelt AL, Sebag-Montefiore D. Phase 2 Neoadjuvant Treatment Intensification Trials in Rectal Cancer: A Systematic Review. Int J Radiat Oncol Biol Phys. 2018 Jan 1;100(1):146-158. doi: 10.1016/j.ijrobp.2017.09.042. Epub 2017 Sep 29. PMID 29254769
- [Background] Caravatta L, Padula GD, Picardi V, Macchia G, Deodato F, Massaccesi M, Sofo L, Pacelli F, Rotondi F, Cecere G, Sallustio G, Di Lullo L, Piscopo A, Mignogna S, Bonomo P, Cellini N, Valentini V, Morganti AG. Concomitant boost radiotherapy and multidrug chemotherapy in the neoadjuvant treatment of locally advanced rectal cancer: results of a phase II study. Acta Oncol. 2011 Nov;50(8):1151-7. doi: 10.3109/0284186X.2011.582880. Epub 2011 Aug 18. PMID 21851185
- [Background] Engels B, Platteaux N, Van den Begin R, Gevaert T, Sermeus A, Storme G, Verellen D, De Ridder M. Preoperative intensity-modulated and image-guided radiotherapy with a simultaneous integrated boost in locally advanced rectal cancer: report on late toxicity and outcome. Radiother Oncol. 2014 Jan;110(1):155-9. doi: 10.1016/j.radonc.2013.10.026. Epub 2013 Nov 12. PMID 24239243
- [Background] Lee JH, Kim DY, Nam TK, Yoon SC, Lee DS, Park JW, Oh JH, Chang HJ, Yoon MS, Jeong JU, Jang HS. Long-term follow-up of preoperative pelvic radiation therapy and concomitant boost irradiation in locally advanced rectal cancer patients: a multi-institutional phase II study (KROG 04-01). Int J Radiat Oncol Biol Phys. 2012 Nov 15;84(4):955-61. doi: 10.1016/j.ijrobp.2012.01.045. Epub 2012 Apr 24. PMID 22537540
- [Background] Li JL, Ji JF, Cai Y, Li XF, Li YH, Wu H, Xu B, Dou FY, Li ZY, Bu ZD, Wu AW, Tham IW. Preoperative concomitant boost intensity-modulated radiotherapy with oral capecitabine in locally advanced mid-low rectal cancer: a phase II trial. Radiother Oncol. 2012 Jan;102(1):4-9. doi: 10.1016/j.radonc.2011.07.030. Epub 2011 Sep 6. PMID 21903285